CLINICAL TRIAL: NCT04817280
Title: Influence of Ice Swimming on Hardening Against SARS-CoV-2 and Influence of AB0 Rh Blood Type on Viral Resistance in Polish Ice Swimmers.
Brief Title: COVID-19 in Polish Ice Swimmers.
Acronym: ICE
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KB-03/139/2021
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Covid19; SARS-CoV Infection; Resistance, Disease; Hypothermia; Hypothermia Due to Cold Environment
Keywords: Ice Swim; Immune System; Immunity; Temporarily cooling down
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Disease Resistance; Hypothermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ice Swimmers Group.: No intervention. Data obtained from Polish ice swimmers reported by them retrospectively in the questionnaire.
  Interventions: Other: Ice Swimming

INTERVENTIONS:
Other: Ice Swimming — The intervention is not made in the course of a research study. Ice swimming has been introduced earlier by a given group. The group was made up of people who already swim in ice.

SUMMARY:
Ice swimming is an increasingly common phenomenon in Poland. It has been confirmed that it has a beneficial effect on health by increasing the natural non-specific immunity to infections. In the face of the current Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) pandemic causing Coronavirus Disease 2019 (COVID-19), researchers decided to use a survey to check the incidence of COVID-19 among Polish ice swimmers, as well as recent ailments. Then, the researchers will compare the obtained results with epidemiological data for Poland.Researchers will also investigate the relationship between susceptibility to SARS-CoV-2 infection and the blood group and Rh factor among ice swimmers.

DETAILED DESCRIPTION:
The research tool is an original questionnaire compiled by a team of experts conducting the study. The survey includes questions about sociodemographic data, such as age and gender and blood type in AB0 system with Rh factor, and questions about the frequency of ice swimming, the duration of a single session, and since when respondents have been ice swimming. There was also a question about the respondents' compliance with the restrictions and recommendations related to the pandemic and contacts with people with confirmed SARS-CoV-2 infection. In the survey, researchers ask about the infectious symptoms experienced during the pandemic and about being diagnosed with COVID-19 or its exclusion. People who have been ill are asked about the place of treatment.

The questionnaires are collected in traditional form, on the Internet and as scans of documents. Each survey was completely anonymous. The obtained statistical data will be compared with official data on new COVID-19 cases and recoveries at the same time. Official data are published by the Ministry of Health and earlier also by Sanitary and Epidemiological Stations. The main aim of the study was to determine whether ice swimming also increases resistance to SARS-CoV-2 and COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* ice swimmers

Exclusion Criteria:

* not active ice swimmers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surveys are distributed en masse among ice swimmers from Poland. Comparative data for the control group is derived from officially published national and regional pandemic data.
Sampling Method: Non-Probability Sample
Enrollment: 2534 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the incidence of COVID-19 among ice swimmers compared to the general population. | 47 days.
  Comparison of the data obtained from surveys collected among ice swimmers with the data published in official channels for the general population during this period.
Assessment of the frequency of asymptomatic SARS-CoV-2 infection among ice swimmers compared to the general population. | 47 days.
  Comparison of the data obtained from surveys collected among ice swimmers with the data published in official channels for the general population during this period.
Assessment of the frequency of occurrence of particular symptoms of SARS-CoV-2 infection among ice swimmers compared to the general population. | 47 days.
  Comparison of the data obtained from surveys collected among ice swimmers with the data published in official channels for the general population during this period.
Assessment of the frequency of COVID-19 treatment in an outpatient, inpatient and intensive care unit among ice swimmers compared to the general population. | 47 days.
  Comparison of the data obtained from surveys collected among ice swimmers with the data published in official channels for the general population during this period.
Assessment of the impact of parameters and ice swimming strategies on the likelihood of developing COVID-19, the occurrence of individual symptoms of the disease and the severity of its course. | 47 days.
  Inference from data obtained from surveys collected among ice swimmers.
Assessment of the influence of blood group on susceptibility to SARS-CoV-2 infection among ice swimmers. | 47 days.
  Inference from data obtained from surveys collected among ice swimmers.

SECONDARY OUTCOMES:
Assessment of the immunity of the ice swimmer's immune system compared to the general population. | 47 days.
  Comparison of the data obtained from surveys collected among ice swimmers with the data published in official channels for the general population during this period.

CONTACTS AND LOCATIONS:
Overall Officials: Sylwia Sulimiera Michalak, MD, PhD, Study Director — Department of Pharmacology and Toxicology, Medical University of Zielona Gora; Edyta Wolny-Rokicka, MD, PhD, Study Director — Department and Center of Radiotherapy, Multidisciplinary Provincial Hospital in Gorzow Wielkopolski; Andrzej Tukiendorf, Prof., Study Chair — Department of Public Health, Wroclaw Medical University; Lukasz K Wysoczanski, MD, Principal Investigator — Department of Family Medicine, Wroclaw Medical University; Paulina N Wysoczanska, MD, Principal Investigator — Department of Family Medicine, Wroclaw Medical University
Locations (3):
- Poland (3):
  - Department of Public Health at Wroclaw Medical University, Wroclaw, Dolny Slask
  - Department of Radiotherapy of Multidisciplinary Provincial Hospital, Gorzów Wielkopolski, Lubusz Voivodeship
  - Treasury Medical Company, Zielona Góra, Lubusz Voivodeship

IPD SHARING:
Plan to Share IPD: No